CLINICAL TRIAL: NCT03847545
Title: Muscle Strain in Multiple Sclerosis Patients Measured by Ultrasound Speckle Tracking
Brief Title: Muscle Strain in Multiple Sclerosis Patients Measured by Ultrasound Speckle Tracking Technique
Acronym: MUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Sygehus Lillebaelt (Other); Region of Southern Denmark (Other); The Augustinus Foundation, Denmark. (Other); Lounkær Fonden (Unknown); Fonden for scleroseramte på Fyn (Unknown); The Danish Multiple Sclerosis Society (Unknown); TH MAIGAARDS EFTF. FRU LILY BENTHINE LUNDS FOND AF 1. JUNI 1978 (Unknown); Fonden til Lægevidenskabens Fremme (Other); Overlægeråds forskningsfond (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mariathorning
Record Dates: First submitted 2018-12-19; First posted 2019-02-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
Keywords: Speckle tracking ultrasonography; Muscle strain; Fampridine; Multiple Sclerosis; Neurological diseases; Biomarkers; muscle contractility
MeSH Terms: conditions — Multiple Sclerosis; Sprains and Strains | interventions — 4-Aminopyridine

STUDY DESIGN:
Intervention Model Description: Prospective cohort Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The participants receive Fampridine treatment (10 mg x 2 daily) for 14 days. They are testet prior to treatment and following the 14 days of treatment.
  Interventions: Drug: Fampridine

INTERVENTIONS:
Drug: Fampridine — sustained-release tablet 10 mg morning and evening.

SUMMARY:
The primary study, as outlined in the original trial registration, aiming to use ultrasound speckle tracking (STU) to monitor muscle contractility in multiple sclerosis (MS) patients receiving vs. not receiving fampridine, as well as to relate these results to performance-based measures and biomarkers to explore disease progression and muscle activity, has been cancelled. Instead four exploratory studies that originate from the initial trial registration but with revised aims, outcome measures and time points, have been prepared - see the DEVIATIONS TO TRIAL PROTOCOL included in the Statistical Analysis Plan filed under "Document section".

Summary of original trial registration:

Despite effective treatments, the majority of patients with multiple sclerosis experience walking impairments to a degree where walking aids or a wheelchair is required. Since 2009, medical treatment of walking impairments has been possible with fampridine, which has proven effective in approximately 40% of the patients. At present, the treatment is offered on the basis of a measurable improved walking function evaluated by simple performance-based walking tests. The treatment is offered on the basis of a measurable improved walking distance.

This is shown today using simple performance-based walking tests that are difficult to complete for those MS patients who are without gait function but could still benefit from fampridine treatment.

Ultrasound speckle tracking is a non-invasive ultrasound technique, with the potential to measure muscle function, including muscle contractility (through strain). Ultrasound speckle tracking is designed for dynamic cardiac muscular examination, but can in a modified version be used for assessment of the skeletal muscles.

The purpose of this project is to use ultrasound speckle tracking to monitor muscle contractility in MS patients receiving vs. not receiving fampridine treatment. Furthermore, to relate these results to biomarkers in blood and urine to examine disease progression and muscle activity.

DETAILED DESCRIPTION:
The primary study, as outlined in the original trial registration, aiming to use ultrasound speckle tracking (STU) to monitor muscle contractility in multiple sclerosis (MS) patients receiving vs. not receiving fampridine, as well as to relate these results to performance-based measures and biomarkers to explore disease progression and muscle activity, has been cancelled. Instead four exploratory studies that originate from the initial trial registration but with revised aims, outcome measures and time points, have been prepared - see the DEVIATIONS TO TRIAL PROTOCOL included in the Statistical Analysis Plan filed under "Document section"

The detailed description that was included in the original trial registration:

Despite effective treatments, the majority of multiple sclerosis (MS) patients experience difficulty in walking and the need of a walker or wheelchair. Since 2009, medical treatment of walking impairments has been possible with fampridine, which has proven effective at approximately 40% of patients.

At present, the treatment is offered on the basis of a measurable improved walking function evaluated by simple performance-based walking tests. Multiple sclerosis patients, who do not have the sufficient gait function to complete these tests, may still benefit from fampridine treatment in other activities of daily life. However, these patients are currently not eligible for fampridine treatment due to current requirements of a measurable improved effect.

Ultrasound speckle tracking (UST) is a non-invasive ultrasound technique, with the potential to directly analyze the muscle strain in the muscles. UST is designed for dynamic cardiac muscular examination, but can be used in a modified version for skeletal muscle examination. The technique has already been tested in a minor pilot study with MS patients.

The objective of the present study is to use UST to monitor muscle strain in the weight-bearing and transfer-related muscles in MS patients who receive fampridine vs. patients who do not receive this treatment. Strain is evaluated over time during different isometric contractions. Furthermore, the relation between these results and the performance based measures of clinical function and biomarkers in blood and urine will be examined to explore disease progression and muscle activity.

MS patients will be recruited from sclerosis clinics at Odense University Hospital (OUH), Esbjerg, Kolding and Sønderborg. All participants will undergo the existing standard practice for patients receiving fampridine treatment, including functional and neurological examination. In addition to the regular practice, participants will be offered UST, answer relevant questionnaires as well as the collection of blood- and urine samples (8 ml of blood and 10 ml of urine will be centrifuged and kept in 0.5 ml aliquots and stored in the already established biobank at the Department of Neurology, OUH.

Participants will be tested at baseline (just before start of fampridine treatment), after 14 days of treatment and again one year after baseline. All three test sessions will include the above mentioned testing protocol. The primary end-point will be at one-year follow-up.

A sub-group of 30 randomly selected participants will supplementary perform a 3-dimensional gait analysis in the motion laboratory. A list generated from 30 randomly found numbers from 1 to 60 will be used. In the motion laboratory, the outcomes: Kinematics, kinetics, gait summary measures and temporo spatial outcome measures will be generated.

Participants, who respond to the fampridine after 14 days of treatment, will continue in the project as cases, whereas non-responders persist in the trial as an untreated control group.

The study is approved by the Regional Committees on Health Research Ethics for Southern Denmark, project Identification: S-20170203. Sample size is based on previously published studies regarding effect of fampridine treatment as well as already detected differences in pilot data obtained from 2 MS patients and 4 healthy controls on m supraspinatus at 40% of maximal load. With an alpha value of p<0.05 and a power of 0.80, sample size is 60.

The study will be conducted in accordance to the Good Clinical Practice and the Declaration of Helsinki and has been approved by the National Committee on Health Research Ethics and the Danish Data Protection Agency.

To our knowledge, this is the first study to evaluate muscle function in MS patients through muscle strain measured using UST as well as examine its correlation to biomarkers for disease progression and muscle activity. Consequently, the result of the present study could expand clinical guidelines for fampridine treatment in MS patients. Furthermore, UST could be implemented for clinical use in assessing muscle strength and treatment response and can ultimately be used to monitor disease progression in MS patients independent of fampridine treatment. The included analysis of blood and urine opens new opportunities for diagnostic and prognostic biomarkers. In addition to provide new knowledge of disease mechanisms, it may also serve as potential new targets for future treatments.

ELIGIBILITY:
Inclusion Criteria:

* Fills the criteria for fampridine treatment
* Fills the diagnostic McDonald criteria for MS
* Age between 18 and 100 years
* EDSS between 4 and 7

Exclusion Criteria:

* Diagnosed epilepsy
* MS attack or an acute decrease of functional capacity within the last 60 days
* Change in immunomodulatory treatment within the last 60 days
* Cancer within the last 5 years
* Clinically significant systemic disease
* Concurrent treatment with cimetidine, carvediol, propanolol and metformine

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Gait Profile Score (GPS) - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in GPS. GPS is a summary measure of kinematic data. The GPS evaluates the overall quality of gait by comparing nine kinematic variables, described as Gait Variable Scores (GVS), relative to normative data.
  GPS is the root mean square (RMS) difference between the data of relevant kinematic variables of an individual patient and the averaged data from a reference group comprised of people without gait impairments.
  Originally we had registred that we would use the Gait Deviation Index (GDI). GDI is a unitless value from 0 to 100. It is based upon kinematic data and is an overall quantitative index that summarises the overall gait pathology into a single score for each patient by comparison with non-pathological gait.
  The GDI and GPS is highly correlated. We chose to use the GPS due to the inclusion of the GVS.

SECONDARY OUTCOMES:
Gait Variable Scores (GVS) - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in GVS. GVS refers to the Root Mean Square difference between the data of the following kinematic variables of an individual patient and the averaged data from a reference group comprised of people without gait impairments:
  Pelvic tilt, obliquity and rotation; hip flexion-extension, adduction-abduction, and rotation; knee flexion-extension; ankle dorsiflexion; and foot progression.
Functional test - 6 Spot Step Test (SSST) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in time it takes the participant to walk through a rectangular area of 1x 5 meters while 5 cylinder blocks must be kicked out of 5 circles marked on the floor.
Functional test - Timed 25 Footwalk (T25-FW) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in time it takes the participant to walk as safe and as quickly as possible through a straight clearly marked lane of 7.62 meters (25 feet).
Functional test - 2-minute Walk Test (2MWT) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in distance that the participant is able to walk in 2 minutes.
Walking speed - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in walking speed (m/s)
Step length - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in step length (m)
Step width - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in step width (m)
Stride length - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in stride length (m)
Cadence - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in cadence (steps/min.)
Questionnaire - 12-Item Multiple Sclerosis Walking Scale (MSWS-12), Danish version | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in MSWS-12. Data is converted to a scale from 0 to 100, where 0 represents the best and 100 the worst. A change score of at least -4 represents a clinically meaningful improvement in the gait function.

OTHER OUTCOMES:
Neurological examination - Expanded Disability Status Scale (EDSS) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in EDSS. The scale ranges from 0 to 10, where 0 indicates that the patient is unaffected by the disease, while 10 indicates death by MS.
Neurological examination - Multiple Sclerosis Impairment Scale (MSIS) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in MSIS. Normal examination corresponds to the value 0 and the theoretical maximum score is 204.
Functional test - Nine Hole Peg Test (9HPT) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in time it takes the participant to collect 9 sticks individually by hand and put them in 9 holes and then to remove them again. The test is performed with each hand.
Peak range of motion (kinematic) - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (follow-up from baseline), 52 weeks (follow-up from "baseline" and "14 days")
  Change in peak range of motion (degrees) for ankle, knee and hip in sagittal, frontal and transverse plane. Measures are captured during a 3D Vicon gait analysis.
Peak and mean joint moments (kinetic) - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in peak and mean joint moments (Nm · BW-1) for ankle, knee and hip in sagittal, frontal and transverse plane. Measures are captured during a 3D Vicon gait analysis. relevant kinetic measures using a 3D Vicon motion capture analysis.
Single support - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in single support (percentage of stride)
Single Limp Index - (subgroup of 30 allocated to 3D gait analysis) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change Limp Index (left vs. right in %)
Questionnaire - Oxford Shoulder Score (OSS), Danish version | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in OSS. Symptoms are rated between 1 (minimal symptoms) and 5 (severe symptoms). The total score of the 12 questions combined is minimum 12 and maximum 60.
Questionnaire - UCLA Activity Scale, Danish version | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in the University of California Los Angeles activity-level rating (UCLA activity scale), Danish version. On a 10-point scale, the option is marked that matches the level of intensity and frequency of physical activity best, where 1 ="Wholly inactive: depend on others, cannot leave residence, and 10 =" Regularly participates in impact sports".
Neurofilament light | Baseline, 14 days (follow-up from baseline), 52 weeks (follow-up from "baseline" and "14 days")
  Change in neurofilament light- biomarker for neurodegeneration. Simoa ELISA in serum/plasma pg/ml
TNF | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in TNF - biomarker for inflammation, ELISA in plasma/serum pg/ml
TNFR1 | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in TNFR1 - biomarker for inflammation, ELISA in plasma/serum pg/ml
TNFR2 | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in TNFR2 - biomarker for inflammation, ELISA in plasma/serum pg/ml
IL-1alpha | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in IL-1alpha, biomarker for inflammation, ELISA in plasma/serum pg/ml
IL-1beta | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in IL-1beta - biomarker for inflammation, ELISA in plasma/serum pg/ml
IL-1Ra | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in IL-1Ra - biomarker for inflammation, ELISA in plasma/serum pg/ml
Creatinin phosphokinase | Baseline, 14 days (follow-up from baseline), 52 weeks (follow-up from "baseline" and "14 days")
  Change in Creatinin phosphokinase - biomarker for muscle function, Enzymassay in plasma/serum micromol/L
Lactate dehydrogenase | Baseline, 14 days (follow-up from baseline), 52 weeks (follow-up from "baseline" and "14 days")
  Change in Lactate dehydrogenase - biomarker for muscle function, Enzymassay Plasma U/liter
Myoglobin | Baseline, 14 days (follow-up from baseline), 52 weeks (follow-up from "baseline" and "14 days")
  Change in myoglobin - biomarker for muscle function, ELISA in urine and plasma microg/L
Skeletal troponin | Baseline, 14 days (follow-up from baseline), 52 weeks (follow-up from "baseline" and "14 days")
  Change in Skeletal troponin - biomarker for muscle function, ELISA in serum/plasma microg/L
eGFR | Baseline, 14 days (follow-up from baseline), 52 weeks (follow-up from "baseline" and "14 days")
  Change in eGFR - biomarker for kidney function, serum/plasma ml/min.
Test for urinary tract infection (UTI) | Baseline, 14 days follow-up, 52 weeks follow-up
  Testing for UTI - marker for infection, using strips
Muscle strain of the supraspinatus muscle | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in muscle strain (percentage of deformation during a contractile cycle of the muscle) before and during fampridine treatment. The muscle strain will be measured during submaximal isometric contractions of 40%, 60% and 80%.
Muscle strain of the biceps brachii muscle | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in muscle strain (percentage of deformation during a contractile cycle of the muscle) before and during fampridine treatment. The muscle strain will be measured during submaximal isometric contractions of 20% 40% and 60%.
Muscle strain of the soleus muscle | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in muscle strain (percentage of deformation during a contractile cycle of the muscle) before and during fampridine treatment. The muscle strain will be measured during submaximal isometric contractions of 20% 40% and 60%.
IL-2 | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in IL-2 - biomarker for inflammation, ELISA in plasma/serum pg/ml
IL-4 | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in IL-4 - biomarker for inflammation, ELISA in plasma/serum pg/ml
IL-8 | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in IL-8 - biomarker for inflammation, ELISA in plasma/serum pg/ml
IL-17 | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in IL-17 - biomarker for inflammation, ELISA in plasma/serum pg/ml
INF-gamma | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in INF-gamma - ELISA in plasma/serum pg/ml
Glial fibrillary acidic protein (GFAP) | Baseline, 14 days (Change from baseline to 14 days follow-up)
  Change in Glial fibrillary acidic protein - biomarker for neurodegeneration. Simoa ELISA in serum/plasma pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Helle H. Nielsen, MD, PhD, Study Director — Department of Neurology, Odense University Hospital, Odense, Denmark; Maria Thorning, MSc, Principal Investigator — Department of Neurology, Odense University Hospital, Odense, Denmark
Locations (1):
- University of Southern Denmark - Odense Univarsity Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become availerble six months after submission. Time period of five years.
Access Criteria: All data are hosted at OPEN (Odense Patient Explorative Network), which allows data sharing upon request.
URL: https://www.sdu.dk/en/om_sdu/institutter_centre/klinisk_institut/forskning/forskningsenheder/open.aspx

REFERENCES:
- [Background] Gottberg K, Einarsson U, Ytterberg C, de Pedro Cuesta J, Fredrikson S, von Koch L, Widen Holmqvist L. Health-related quality of life in a population-based sample of people with multiple sclerosis in Stockholm County. Mult Scler. 2006 Oct;12(5):605-12. doi: 10.1177/1352458505070660. PMID 17086907
- [Background] Goodman AD, Brown TR, Edwards KR, Krupp LB, Schapiro RT, Cohen R, Marinucci LN, Blight AR; MSF204 Investigators. A phase 3 trial of extended release oral dalfampridine in multiple sclerosis. Ann Neurol. 2010 Oct;68(4):494-502. doi: 10.1002/ana.22240. PMID 20976768
- [Background] Goodman AD, Brown TR, Krupp LB, Schapiro RT, Schwid SR, Cohen R, Marinucci LN, Blight AR; Fampridine MS-F203 Investigators. Sustained-release oral fampridine in multiple sclerosis: a randomised, double-blind, controlled trial. Lancet. 2009 Feb 28;373(9665):732-8. doi: 10.1016/S0140-6736(09)60442-6. PMID 19249634
- [Background] Solari A, Uitdehaag B, Giuliani G, Pucci E, Taus C. Aminopyridines for symptomatic treatment in multiple sclerosis. Cochrane Database Syst Rev. 2001;2002(4):CD001330. doi: 10.1002/14651858.CD001330. PMID 11687106
- [Background] Jensen H, Ravnborg M, Mamoei S, Dalgas U, Stenager E. Changes in cognition, arm function and lower body function after slow-release Fampridine treatment. Mult Scler. 2014 Dec;20(14):1872-80. doi: 10.1177/1352458514533844. Epub 2014 May 22. PMID 24852920
- [Background] Jensen HB, Mamoei S, Ravnborg M, Dalgas U, Stenager E. Distribution-based estimates of minimum clinically important difference in cognition, arm function and lower body function after slow release-fampridine treatment of patients with multiple sclerosis. Mult Scler Relat Disord. 2016 May;7:58-60. doi: 10.1016/j.msard.2016.03.007. Epub 2016 Mar 18. PMID 27237758
- [Background] Jensen HB, Ravnborg M, Dalgas U, Stenager E. 4-Aminopyridine for symptomatic treatment of multiple sclerosis: a systematic review. Ther Adv Neurol Disord. 2014 Mar;7(2):97-113. doi: 10.1177/1756285613512712. PMID 24587826
- [Background] Mondillo S, Galderisi M, Mele D, Cameli M, Lomoriello VS, Zaca V, Ballo P, D'Andrea A, Muraru D, Losi M, Agricola E, D'Errico A, Buralli S, Sciomer S, Nistri S, Badano L; Echocardiography Study Group Of The Italian Society Of Cardiology (Rome, Italy). Speckle-tracking echocardiography: a new technique for assessing myocardial function. J Ultrasound Med. 2011 Jan;30(1):71-83. doi: 10.7863/jum.2011.30.1.71. PMID 21193707
- [Background] Frich, L.H., et al., Direct isometric muscle strain analyses using speckle tracking technology. A validation study, in European Muscle Conference 2017. 2017, Journal of Muscle Research and Cell Motility: Potsdam
- [Derived] Thorning M, Nielsen HH, Frich LH, Jensen HB, Lambertsen KL, Holsgaard-Larsen A. Gait quality and function after fampridine treatment in patients with multiple sclerosis - A prospective cohort study. Clin Biomech (Bristol). 2022 Dec;100:105826. doi: 10.1016/j.clinbiomech.2022.105826. Epub 2022 Nov 17. PMID 36436320

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT03847545/SAP_000.pdf
  • Informed Consent Form (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT03847545/ICF_001.pdf